CLINICAL TRIAL: NCT05066919
Title: Operative Versus Non-operative Treatment of Recalcitrant Plantar Fasciitis - A Randomized Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to local changes in patient up-take after COVID it is no longer possible to conduct the study.
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Christopher Jantzen, MD., Principal Investigator, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 78652
Record Dates: First submitted 2021-09-30; First posted 2021-10-04 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Plantar Fascitis; Surgical Treatment; Non-operative Treatment; Randomized Study
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative treatment (Experimental): Patients treated with open plantar fasciotomy
  Interventions: Procedure: Open plantar fasciotomy
- Conservative treatment (Active Comparator): Patients treated non-operatively with exercise
  Interventions: Other: Conservative treatment

INTERVENTIONS:
Procedure: Open plantar fasciotomy — In the surgical treated group, the plantar fascia is defined percutaneously (medial and lateral margin). An incision is then made just distal to the heel pad medially over the plantar fascia. A resection is performed 1 cm in length with a width corresponding to 50% of the medial band. The skin is sutured with nylon/nonresorbable suture. Postoperatively, the operated foot is elevated for the first 24 hours. Then free mobilization in postoperative shoe (ProCare shoe) is allowed. The dressing is left untouched for 3-5 days, after which it can be changed to a patch. After 14 days the sutures are removed and the patient allowed using regular shoes.
  Arms: Operative treatment
Other: Conservative treatment — In the conservative treatment group, patients are instructed in performing stretching exercises with plantar fascia specific stretching exercises 10 x 10 seconds, 3 times daily and high load strength training are every other day for 3 months. Each high load strength exercise consists of 3 seconds of concentric phase (lifting up with the heel) and 3 seconds of eccentric phase (lowering the heel) with 2 seconds of isometric pause (pause at maximum lifted heel). 12 repetitions max (RM) are performed, defined as the maximum (over) weight the patient can lift 12 times with full range of motion while performing the exercise correctly. 3 x 12 exercises are performed per workout. After 2 weeks, the load is while the number of repetitions is reduced to 10 RM with an increase to 4 repetitions per workout. After 4 weeks the intensity is increased to 8RM with 5 set. Patients are instructed to increase the load throughout the training period.
  Arms: Conservative treatment

SUMMARY:
The purpose of the study is to examine whether patients with heel spurs for more than 6 months, who have been treated conservatively, have better effect of surgery than further conservative treatment. The study is performed as a randomized trial with the inclusion of 32 patients divided between open plantar fasciectomy and conservative treatment.

The primary endpoint is Self-Reported-Foot-And-Ankle Score (SEFAS-score) after 24 months.

Secondary endpoints includes: Pain (Visual analogue score) at first step, rest and activity after 3, 6, 12 and 24 months, SEFAS-score after 3, 6 og 12 months, changes in gait after 6 months (measured with gait-analysis). All endpoints are measured at inclusion.

The power calculation is based on the assumption that surgical treatment gives an improvement in SEFAS-score of 10 points (SD 7.9) after 24 months when compared to conservative treatment together with an alpha-value of 5 % and a beta value of 90 %.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Isolated plantar fasciitis through more than 6 months
* Ultrasonic verification of diagnosis (plantar fascia >4 mm)
* Ability to follow the post-operative- and conservative plans
* Able to give informed consent.

Exclusion Criteria:

* Previous surgical treatment of plantar fasciitis or surgery around the heel
* Rheumatic disease
* Diabetes
* Dementia
* Neuropathy
* Known alcohol abuse
* Pareses/paralysis of the affected extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Self-Reported-Foot-And-Ankle Score (SEFAS) | 24 Months
  The questionnaire contains 12 items with 5 response options. The questionnaire covers different constructs, which are not reported separately in subscales. The most important of these constructs are pain, function, and limitation of function. Each of the 12 multiple-choice questions scores from 0 to 4 where a sum of 0 points represents the most severe disability and 48 represents normal function.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Department of Ortopedic Surgery, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No